CLINICAL TRIAL: NCT04325243
Title: Efficacy of Sildenafil Citrate to Reduce the Rate of Cesarean Section for Intrapartum Fetal Distress During Induction of Labor
Brief Title: Sildenafil Citrate and Intrapartum Fetal Distress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SC-IPFD
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 50 mg oral sildenafil citrate tablet
  Interventions: Drug: Sildenafil 50 mg
- placebo group (Placebo Comparator): placebo tablets of the same shape, color and size of sildenafil citrate tablets
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Sildenafil 50 mg — 50 mg oral Sildenafil tablet
  Arms: study group
Drug: Placebo oral tablet — placebo tablets of the same shape, color and size of Sildenafil tablets manufactured in the Department of Pharmaceuticals, Faculty of Pharmacy
  Arms: placebo group

SUMMARY:
Induction of labour (IOL) is done for 20% of pregnancies for various maternal and fetal indications and nearly 20% of labour inductions end up in caesarean section. The most common causes are failed induction and intrapartum fetal distress. In spite of significant advances in methods of IOL and intrapartum fetal monitoring, no interventions are proven to reduce the development of intrapartum fetal distress

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Pregnant ≥ 37 weeks gestation.
3. Fetus with longitudinal lie and vertex presentation.
4. Healthy fetus with EFW>2500 gm

Exclusion Criteria:

1. Patients with previous cesarean delivery or uterine surgery.
2. Antepartum hemorrhage.
3. Cephalopelvic disproportion.
4. Category II or III non-stress test.
5. Medical disease as hypertension, cardiac, renal and hepatic disorders
6. Intrauterine fetal death.
7. Fetal growth restriction.
8. Fetuses with major congenital malformations.
9. Women taking any anti-hypertensive medication, alpha-adrenergic blocking agents, calcium channel blockers (verapamil), nitrates, medications used to treat pulmonary arterial hypertension, and other phosphodiesterase type 5 inhibitors.
10. Women with a contra-indication to sildenafil treatment such as hypersensitivity to sildenafil.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The rate of cesarean section for intrapartum fetal distress | 24 hours
  Fetus will be considered to be distressed if Ominous fetal heart rate changes led to cesarean section was present

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt